CLINICAL TRIAL: NCT02808312
Title: A Phase 1 Open-Label, Parallel-Group, Adaptive, Single-Dose Study to Evaluate the Pharmacokinetics and Pharmacodynamics of GS-9674 in Subjects With Normal and Impaired Hepatic Function
Brief Title: Pharmacokinetics and Pharmacodynamics of Cilofexor in Adults With Normal and Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-402-3885
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Nonalcoholic Steatohepatitis (NASH); Primary Sclerosing Cholangitis (PSC)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Cholangitis, Sclerosing | interventions — cilofexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment will receive a single oral dose of cilofexor 30 mg (3 x 10 mg tablets).
  Interventions: Drug: Cilofexor
- Cohort 1: Normal Hepatic Function (Experimental): Matched normal hepatic function participants to mild hepatic impairment participants will receive a single oral dose of cilofexor 30 mg (3 x 10 mg tablets).
  Interventions: Drug: Cilofexor
- Cohort 2: Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment will receive a single oral dose of cilofexor 30 mg (3 x 10 mg tablets).
  Interventions: Drug: Cilofexor
- Cohort 2: Normal Hepatic Function (Experimental): Matched normal hepatic function participants to moderate hepatic impairment participants will receive a single oral dose of cilofexor 30 mg (3 x 10 mg tablets).
  Interventions: Drug: Cilofexor
- Cohort 3: Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment will receive a single oral dose of cilofexor 10 mg (1 x 10 mg tablet).
  Interventions: Drug: Cilofexor
- Cohort 3: Normal Hepatic Function (Experimental): Matched normal hepatic function participants to severe hepatic impairment participants will receive a single oral dose of cilofexor 10 mg (1 x 10 mg tablet).
  Interventions: Drug: Cilofexor

INTERVENTIONS:
Drug: Cilofexor — Tablet(s) administered orally in a fed state on Day 1
  Other Names: GS-9674

SUMMARY:
The primary objective of this study is to evaluate the single-dose pharmacokinetics of cilofexor in adults with impaired hepatic function relative to matched, healthy controls with normal hepatic function.

ELIGIBILITY:
Key Inclusion Criteria:

Cohort 1:

* Individuals with mildly impaired and normal hepatic function.
* Individuals with mild hepatic impairment must have a score of 5-6 on the Child-Pugh-Turcotte (CPT) classification at screening without evidence of worsening clinical and/or laboratory signs of hepatic impairment within 2 months prior or within the screening period.

Cohort 2:

* Individuals with moderately impaired and normal hepatic function.
* Individuals with moderate hepatic impairment must have a score of 7-9 on the CPT classification at screening without evidence of worsening clinical and/or laboratory signs of hepatic impairment within 2 months prior or within the screening period.

Cohort 3:

* Individuals with severely impaired and normal hepatic function.
* Individuals with severe hepatic impairment must have a score of 10-15 on the CPT classification at screening without evidence of worsening clinical and/or laboratory signs of hepatic impairment within 2 months prior or within the screening period.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- United States (4):
  - Miami, Florida
  - Orlando, Florida
  - Knoxville, Tennessee
  - San Antonio, Texas
- Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States (US) and New Zealand. The first participant was screened on 13 July 2016. The last study visit occurred on 16 October 2018.
Pre-assignment Details: In the control groups (normal hepatic function), each participant was matched for age, gender, race, and body mass index with a participant in the hepatic impairment group. 17 total unique participants with normal hepatic function were enrolled in Cohort 1 (N = 10) and Cohort 2 (N = 7). 5 participants with normal hepatic function from Cohort 1 also served as matched controls in Cohort 2.
Groups:
- Cohort 1: Mild Hepatic Impairment: Participants with mild hepatic impairment received a single oral dose of cilofexor 30 mg (3 x 10 mg tablets) in a fed state, on Day 1.
- Cohort 2: Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single oral dose of cilofexor 30 mg (3 x 10 mg tablets) in a fed state, on Day 1.
- Cohort 1 & 2: Normal Hepatic Function: Matched normal hepatic function participants to mild or moderate hepatic impairment participants received a single oral dose of cilofexor 30 mg (3 x 10 mg tablets) in a fed state, on Day 1.
- Cohort 3: Severe Hepatic Impairment: Participants with severe hepatic impairment received a single oral dose of cilofexor 10 mg (1 x 10 mg tablet) in a fed state, on Day 1.
- Cohort 3: Normal Hepatic Function: Matched normal hepatic function participants to severe hepatic impairment participants, received a single oral dose of cilofexor 10 mg (1 x 10 mg tablet) in a fed state, on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 2: Moderate Hepatic Impairment | Cohort 1 & 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Started | 10 | 10 | 17 | 10 | 10
Completed | 10 | 10 | 16 | 10 | 10
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Enrolled but Never Treated | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Cohort 1 & 2: Normal Hepatic Function: Matched normal hepatic function participants to mild or moderate hepatic impairment participants, received a single oral dose of cilofexor 30 mg (3 x 10 mg tablets) in a fed state, on Day 1.
- Cohort 3: Normal Hepatic Function: Matched normal hepatic function participants, received a single oral dose of cilofexor 30 mg (3 x 10 mg tablets ) or 10 mg (1 x 10 mg tablet) in a fed state, on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 2: Moderate Hepatic Impairment | Cohort 1 & 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function | Total
Number analyzed (Participants) | 10 | 10 | 16 | 10 | 10 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10.1) | 57 (8.9) | 55 (7.6) | 54 (9.5) | 52 (8.4) | 54.45 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5 | 3 | 3 | 16
  Male | 7 | 8 | 11 | 7 | 7 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7 | 6 | 5 | 25
  Not Hispanic or Latino | 6 | 7 | 9 | 4 | 5 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 1 | 3
  White | 8 | 10 | 15 | 9 | 9 | 51
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 2 | 1 | 3 | 1 | 1 | 8
  United States | 8 | 9 | 13 | 9 | 9 | 48

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUClast of Cilofexor
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: ≤ 5 minutes predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, and 96 hours postdose on Day 1
Population: The PK Analysis Sets included all enrolled participants who took at least 1 dose of study drug and had at least 1 nonmissing postdose concentration value reported by the PK laboratory for the corresponding analytes. A participant with normal hepatic function might serve as a matched control across cohorts evaluating the same cilofexor dose.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Cohort 1: Normal Hepatic Function: Matched normal hepatic function participants to mild hepatic impairment participants, received a single oral dose of cilofexor 30 mg (3 x 10 mg tablets) in a fed state, on Day 1.
- Cohort 2: Normal Hepatic Function: Matched normal hepatic function participants to moderate hepatic impairment participants, received a single oral dose of cilofexor 30 mg (3 x 10 mg tablets) in a fed state, on Day 1.
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
h*ng/mL | 5381.0 (2175.34) | 2972.6 (1230.49) | 8223.7 (7492.41) | 2756.7 (851.38) | 6534.3 (3791.05) | 960.0 (352.71)
Statistical Analysis 1: Comparison: Cohort 1: Mild Hepatic Impairment vs Cohort 1: Normal Hepatic Function; An analysis of variance (ANOVA) model with hepatic function group as a fixed effect was fitted to the natural logarithmic transformation of PK parameters (AUClast) for each cohort; Test type: Other — Two-sided 90% Confidence Intervals (CIs) were calculated for the ratios of geometric least-squares means (GLSMs) of PK parameters between mild hepatic impairment group and the control (normal hepatic function) group; GLSM ratio = 1.7869, 90% CI 2-sided [1.2885 to 2.4781]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Hepatic Impairment vs Cohort 2: Normal Hepatic Function; An ANOVA model with hepatic function group as a fixed effect was fitted to the natural logarithmic transformation of PK parameters (AUClast) for each cohort; Test type: Other — Two-sided 90% CIs were calculated for the ratios of GLSMs of PK parameters between moderate hepatic impairment group and the control (normal hepatic function) group; GLSM ratio = 2.4868, 90% CI 2-sided [1.6735 to 3.6954]
Statistical Analysis 3: Comparison: Cohort 3: Severe Hepatic Impairment vs Cohort 3: Normal Hepatic Function; [analysis description as in outcome 1, analysis 2]; Test type: Other — Two-sided 90% CIs were calculated for the ratios of GLSMs of PK parameters between severe hepatic impairment group and the control (normal hepatic function) group; GLSM ratio = 6.3240, 90% CI 2-sided [4.3675 to 9.1569]

2. Primary Outcome: PK Parameter: AUCinf of Cilofexor
Description: AUCinf is defined as the concentration of drug extrapolated to infinite time.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed. A participant with normal hepatic function might serve as a matched control across cohorts evaluating the same cilofexor dose.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
h*ng/mL | 5411.9 (2181.82) | 3024.3 (1224.02) | 8288.2 (7583.42) | 2805.6 (851.26) | 6719.4 (4056.73) | 986.2 (354.93)
Statistical Analysis 1: Comparison: Cohort 1: Mild Hepatic Impairment vs Cohort 1: Normal Hepatic Function; An ANOVA model with hepatic function group as a fixed effect was fitted to the natural logarithmic transformation of PK parameters (AUCinf) for each cohort; Test type: Other — Two-sided 90% CIs were calculated for the ratios of GLSMs of PK parameters between mild hepatic impairment group and the control (normal hepatic function) group; GLSM ratio = 1.7628, 90% CI 2-sided [1.2750 to 2.4374]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Hepatic Impairment vs Cohort 2: Normal Hepatic Function; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; GLSM ratio = 2.4559, 90% CI 2-sided [1.6531 to 3.6486]
Statistical Analysis 3: Comparison: Cohort 3: Severe Hepatic Impairment vs Cohort 3: Normal Hepatic Function; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 3]; GLSM ratio = 6.2497, 90% CI 2-sided [4.2965 to 9.0910]

3. Primary Outcome: PK Parameter: Cmax of Cilofexor
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
ng/mL | 994.1 (533.38) | 603.5 (275.33) | 909.2 (477.20) | 495.7 (199.45) | 426.6 (136.40) | 182.4 (86.67)
Statistical Analysis 1: Comparison: Cohort 1: Mild Hepatic Impairment vs Cohort 1: Normal Hepatic Function; An ANOVA model with hepatic function group as a fixed effect was fitted to the natural logarithmic transformation of PK parameters (Cmax) for each cohort; Test type: Other — [test comment as in outcome 2, analysis 1]; GLSM ratio = 1.5703, 90% CI 2-sided [1.0723 to 2.2995]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Hepatic Impairment vs Cohort 2: Normal Hepatic Function; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 2]; GLSM ratio = 1.7343, 90% CI 2-sided [1.2193 to 2.4667]
Statistical Analysis 3: Comparison: Cohort 3: Severe Hepatic Impairment vs Cohort 3: Normal Hepatic Function; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 3]; GLSM ratio = 2.5369, 90% CI 2-sided [1.7562 to 3.6648]

4. Primary Outcome: PK Parameter: %AUCexp of Cilofexor
Description: %AUCexp is defined as the percentage of AUC extrapolated between AUClast and AUCinf.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of AUCexp
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
percentage of AUCexp | 0.63 (0.270) | 1.95 (1.621) | 0.64 (0.194) | 1.87 (1.653) | 1.81 (1.874) | 2.96 (1.962)

5. Primary Outcome: PK Parameter: Clast of Cilofexor
Description: Clast is defined as the last observable concentration of drug.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
ng/mL | 1.97 (1.005) | 3.84 (2.162) | 2.76 (3.377) | 3.73 (2.378) | 6.03 (8.044) | 2.18 (1.387)

6. Primary Outcome: PK Parameter: Tmax of Cilofexor
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
hours | 3.75 [2.50 to 5.00] | 3.00 [2.50 to 4.00] | 4.50 [2.50 to 10.00] | 3.75 [2.50 to 4.00] | 5.00 [5.00 to 6.00] | 4.00 [3.00 to 5.00]

7. Primary Outcome: PK Parameter: Tlast of Cilofexor
Description: Tlast is defined as the time (observed time point) of Clast.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
hours | 64.80 [48.00 to 72.02] | 48.00 [24.00 to 72.00] | 72.00 [72.00 to 96.00] | 48.00 [24.00 to 72.00] | 96.00 [96.00 to 96.00] | 48.00 [24.00 to 48.00]

8. Primary Outcome: PK Parameter: λz of Cilofexor
Description: λz is defined as the terminal elimination rate constant, estimated by linear regression of the terminal elimination phase of the log plasma concentration of drug versus time curve of the drug.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
1/hour | 0.070 (0.0377) | 0.099 (0.0661) | 0.051 (0.0152) | 0.100 (0.0655) | 0.045 (0.0117) | 0.099 (0.0659)

9. Primary Outcome: PK Parameter: CL/F of Cilofexor
Description: CL/F is defined as the apparent oral clearance following administration of the drug.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
mL/h | 6621.5 (3219.50) | 11324.4 (4184.32) | 5264.4 (2686.26) | 11631.7 (3666.25) | 1963.1 (964.19) | 11535.9 (4627.39)

10. Primary Outcome: PK Parameter: Vz/F of Cilofexor
Description: Vz/F is defined as the apparent volume of distribution of the drug.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
mL | 97797.6 (18500.74) | 148898.5 (81520.19) | 99541.7 (31192.41) | 153854.9 (83844.37) | 41375.1 (11767.71) | 160423.9 (92259.03)

11. Primary Outcome: PK Parameter: t1/2 of Cilofexor
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
hours | 11.45 [8.50 to 12.94] | 9.49 [4.78 to 11.67] | 13.53 [11.56 to 18.15] | 8.12 [4.90 to 15.02] | 15.90 [12.85 to 19.02] | 9.31 [5.15 to 11.61]

12. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Time Frame: Day 1 up to Day 31
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1 and 2: Normal Hepatic Function: Matched normal hepatic function participants to mild or moderate hepatic impairment participants, received a single oral dose of cilofexor 30 mg (3 x 10 mg tablets) in a fed state, on Day 1.
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 2: Moderate Hepatic Impairment | Cohort 1 and 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 16 | 10 | 10
percentage of participants | 10.0 | 20.0 | 12.5 | 30.0 | 0

13. Secondary Outcome: Percentage of Participants Who Experienced Graded Laboratory Abnormalities
Description: A treatment-emergent laboratory abnormality was defined as an increase of at least 1 toxicity grade from predose at any time postdose up to and including the date of last study drug dose plus 30 days. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: Day 1 up to Day 31
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 2: Moderate Hepatic Impairment | Cohort 1 and 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 16 | 10 | 10
percentage of participants
  Any Laboratory Abnormality | 90.0 | 100.0 | 50.0 | 100.0 | 60.0
  Grade 3 or above Laboratory Abnormalities | 20.0 | 20.0 | 0 | 40.0 | 0

14. Secondary Outcome: Pharmacodynamic (PD) Parameter: Mean Day 1/ Day -1 Ratio of AUC2-12 for α-hydroxy-4-cholesten-3-one (C4)
Description: AUC2-12 is defined as area under the curve calculated by the trapezoidal rule for the time from 2 to 12 hours. For PD assessments on Day -1, participants were administered a single oral dose of placebo-to-match cilofexor tablet on Day -1; the reported Time Frame is with respect to the placebo dosing.
Time Frame: 0.5 hour predose, ≤ 5 minutes predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, and 16 hours postdose on Day -1 and Day 1; 4.5 hours postdose on Day -1; 24, 48, 72, and 96 hours postdose on Day 1
Population: Participants in the PD Analysis Set were analyzed. A participant with normal hepatic function might serve as a matched control across cohorts evaluating the same cilofexor dose.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
ratio | 0.706 (0.2273) | 0.817 (0.2836) | 0.716 (0.2370) | 0.681 (0.2614) | 1.063 (0.2469) | 0.978 (0.4155)
Statistical Analysis 1: Comparison: Cohort 1: Mild Hepatic Impairment vs Cohort 1: Normal Hepatic Function; Test type: Other — Two-sided 90% CIs were calculated for the ratios of GLSMs of PD parameters between mild hepatic impairment group and the control (normal hepatic function) group; GLSM ratio = 0.8722, 90% CI 2-sided [0.6827 to 1.1144]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Hepatic Impairment vs Cohort 2: Normal Hepatic Function; Test type: Other — Two-sided 90% CIs were calculated for the ratios of GLSMs of PD parameters between moderate hepatic impairment group and the control (normal hepatic function) group; GLSM ratio = 1.0731, 90% CI 2-sided [0.8295 to 1.3883]
Statistical Analysis 3: Comparison: Cohort 3: Severe Hepatic Impairment vs Cohort 3: Normal Hepatic Function; Test type: Other — Two-sided 90% CIs were calculated for the ratios of GLSMs of PD parameters between severe hepatic impairment group and the control (normal hepatic function) group; GLSM ratio = 1.1475, 90% CI 2-sided [0.8783 to 1.4992]

15. Secondary Outcome: PD Parameter: Mean Day 1/ Day -1 Ratio of Cmin for α-hydroxy-4-cholesten-3-one (C4)
Description: Cmin for C4 is defined as the minimum observed concentration of C4. For PD assessments on Day -1, participants were administered a single oral dose of placebo-to-match cilofexor tablet on Day -1; the reported Time Frame is with respect to the placebo dosing.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
ratio | 0.599 (0.3272) | 0.707 (0.2838) | 0.668 (0.2384) | 0.583 (0.1634) | 0.953 (0.2073) | 0.727 (0.2674)
Statistical Analysis 1: Comparison: Cohort 1: Mild Hepatic Impairment vs Cohort 1: Normal Hepatic Function; Test type: Other — [test comment as in outcome 14, analysis 1]; GLSM ratio = 0.8188, 90% CI 2-sided [0.5837 to 1.1486]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Hepatic Impairment vs Cohort 2: Normal Hepatic Function; Test type: Other — [test comment as in outcome 14, analysis 2]; GLSM ratio = 1.1323, 90% CI 2-sided [0.8772 to 1.4615]
Statistical Analysis 3: Comparison: Cohort 3: Severe Hepatic Impairment vs Cohort 3: Normal Hepatic Function; Test type: Other — [test comment as in outcome 14, analysis 3]; GLSM ratio = 1.3563, 90% CI 2-sided [1.0468 to 1.7574]

16. Secondary Outcome: PD Parameter: Mean Day 1/ Day -1 Ratio of AUC2-12 for Fibroblast Growth Factor 19 (FGF19)
Description: as for outcome 14
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
ratio | 3.031 (1.0376) | 2.840 (0.9254) | 3.730 (1.3768) | 2.848 (1.0250) | 1.582 (0.8182) | 2.179 (1.6972)
Statistical Analysis 1: Comparison: Cohort 1: Mild Hepatic Impairment vs Cohort 1: Normal Hepatic Function; Test type: Other — [test comment as in outcome 14, analysis 1]; GLSM ratio = 1.0658, 90% CI 2-sided [0.8275 to 1.3726]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Hepatic Impairment vs Cohort 2: Normal Hepatic Function; Test type: Other — [test comment as in outcome 14, analysis 2]; GLSM ratio = 1.2942, 90% CI 2-sided [0.9663 to 1.7334]
Statistical Analysis 3: Comparison: Cohort 3: Severe Hepatic Impairment vs Cohort 3: Normal Hepatic Function; Test type: Other — [test comment as in outcome 14, analysis 3]; GLSM ratio = 0.8225, 90% CI 2-sided [0.5479 to 1.2347]

17. Secondary Outcome: PD Parameter: Mean Day 1/ Day -1 Ratio of Cmax for Fibroblast Growth Factor 19 (FGF19)
Description: Cmax for FGF19 is defined as the maximum observed concentration of FGF19. For PD assessments on Day -1, participants were administered a single oral dose of placebo-to-match cilofexor tablet on Day -1; the reported Time Frame is with respect to the placebo dosing.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 1: Normal Hepatic Function | Cohort 2: Moderate Hepatic Impairment | Cohort 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
ratio | 3.778 (1.4954) | 3.494 (1.4423) | 4.459 (1.9899) | 3.145 (1.4484) | 1.899 (1.1619) | 2.098 (1.1579)
Statistical Analysis 1: Comparison: Cohort 1: Mild Hepatic Impairment vs Cohort 1: Normal Hepatic Function; Test type: Other — [test comment as in outcome 14, analysis 1]; GLSM ratio = 1.0806, 90% CI 2-sided [0.7910 to 1.4762]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Hepatic Impairment vs Cohort 2: Normal Hepatic Function; Test type: Other — [test comment as in outcome 14, analysis 2]; GLSM ratio = 1.3729, 90% CI 2-sided [0.9663 to 1.9506]
Statistical Analysis 3: Comparison: Cohort 3: Severe Hepatic Impairment vs Cohort 3: Normal Hepatic Function; Test type: Other — [test comment as in outcome 14, analysis 3]; GLSM ratio = 0.9030, 90% CI 2-sided [0.6142 to 1.3275]

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 31
Description: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | Cohort 1: Mild Hepatic Impairment | Cohort 2: Moderate Hepatic Impairment | Cohort 1 and 2: Normal Hepatic Function | Cohort 3: Severe Hepatic Impairment | Cohort 3: Normal Hepatic Function
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/16 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/16 | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10 | 2/16 | 2/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Mild Hepatic Impairment (N=10) | Cohort 2: Moderate Hepatic Impairment (N=10) | Cohort 1 and 2: Normal Hepatic Function (N=16) | Cohort 3: Severe Hepatic Impairment (N=10) | Cohort 3: Normal Hepatic Function (N=10)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Mild Hepatic Impairment (N=10) | Cohort 2: Moderate Hepatic Impairment (N=10) | Cohort 1 and 2: Normal Hepatic Function (N=16) | Cohort 3: Severe Hepatic Impairment (N=10) | Cohort 3: Normal Hepatic Function (N=10)
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT02808312/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT02808312/SAP_001.pdf